CLINICAL TRIAL: NCT05124184
Title: Retrospective Post-Market Clinical Follow-Up Study of GORE-TEX® Vascular Grafts and GORE® PROPATEN® Vascular Graft in Peripheral Artery Disease, Aortic Aneurysms, and Dialysis Access
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VGP 21-01
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: PAD - Peripheral Arterial Disease; AAA - Abdominal Aortic Aneurysm; End-Stage Renal Disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- PAD Cohort: Patient was treated for peripheral arterial disease or peripheral arterial aneurysm requiring bypass treated with GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft or GORE® PROPATEN® Vascular Graft
  Interventions: Device: GORE® PROPATEN® Vascular Graft; Device: GORE-TEX® Vascular Grafts
- AAA Cohort: Patient underwent simultaneous or staged aortic aneurysm repair (open surgical AAA or TAAA) involving a GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft
  Interventions: Device: GORE-TEX® Vascular Grafts
- Dialysis Access Cohort: Patient required the creation of a vascular access graft for hemodialysis secondary to a diagnosis of End-Stage Renal Disease using a GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft or GORE® PROPATEN® Vascular Graft
  Interventions: Device: GORE® PROPATEN® Vascular Graft; Device: GORE-TEX® Vascular Grafts

INTERVENTIONS:
Device: GORE® PROPATEN® Vascular Graft — Patients that have had treatment with GORE® PROPATEN® Vascular Graft
  Groups: Dialysis Access Cohort; PAD Cohort
Device: GORE-TEX® Vascular Grafts — Patients that have had treatment with GORE-TEX® Vascular Grafts

SUMMARY:
This multicenter, single-arm retrospective registry (chart review) is being conducted to confirm the clinical performance and safety of GORE-TEX® Vascular Grafts and GORE® PROPATEN® Vascular Graft throughout the device functional lifetime for each indication area.

DETAILED DESCRIPTION:
Up to 9 sites in Europe will be required to enroll 353 patients that have had treatment with GORE-TEX® Vascular Grafts or GORE® PROPATEN® Vascular Grafts in the following indication areas:

144 patients in PAD Cohort

* 72 Patients with any GORE-TEX® Vascular Graft
* 72 Patients with GORE® PROPATEN® 65 patients in Aortic Aneurysm Cohort with GORE-TEX® Vascular Graft 144 patients in Dialysis Access Cohort
* 72 patients implanted with any GORE-TEX® Vascular Graft
* 72 Patients implanted with Patients with GORE® PROPATEN®

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Patient is willing and able to provide written informed consent or consent is waived, according to national and local regulations.
2. Patient was at least 18 years of age at the time of implant.

PAD Cohort Inclusion Criteria 1. Patient was treated for peripheral arterial disease or peripheral arterial aneurysm requiring bypass treated with GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft or GORE® PROPATEN® Vascular Graft at least 5 years before site initiation.

Aortic Aneurysm Cohort Inclusion Criteria

1. Patient underwent simultaneous or staged aortic aneurysm repair (open surgical AAA or TAAA) involving a GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft at least 5 years before site initiation. Research device could have been used to replace or bypass either a diseased visceral branch or the aorta itself.

Dialysis Access Cohort Inclusion Criteria 1. Patient required the creation of a vascular access graft for hemodialysis secondary to a diagnosis of End-Stage Renal Disease using a GORE-TEX® Vascular Graft, GORE® INTERING® Vascular Graft, GORE-TEX® Stretch Vascular Graft or GORE® PROPATEN® Vascular Graft at least 2 years before site initiation with the intent to cannulate the registry device.

Exclusion Criteria:

General Exclusion Criteria

1. Patient was not available for follow up (on-site or remotely) at the clinical site, with the exception of death (e.g., patient lost to follow-up immediately after treatment, patients who live far away from the clinical site and are not available to share follow-up data performed locally).
2. At the time of treatment, patient had known coagulation disorders, including hypercoagulability, that were not amenable to treatment.
3. Patient was pregnant at the time of treatment.
4. Patient had known or suspected systemic infection or infection at the site of graft implantation at the time of implant.
5. Patient had a separate major interventional or surgical vascular procedure within 30 days prior to treatment. CVC catheter placement would be permitted.
6. Patient is already enrolled in this registry under a different cohort.

PAD Cohort Exclusion Criteria

At the time of treatment, the patient must not have met any of the following criteria:

1. Patient had percutaneous transluminal angioplasty (PTA) or stenting of the target artery at the anticipated site of the proximal or distal anastomosis within 30 days prior to the index procedure. Use of PTA or stenting during the index procedure is permitted.
2. Patient had a stroke or myocardial infarction (MI) within 6 weeks prior to the index procedure.
3. Patient has previous instance of Heparin-induced Thrombocytopenia type 2 or has known hypersensitivity to heparin.
4. Patient required composite bypass for index procedure (graft + significant length of autologous vessel). Autologous "cuffs" or patches are allowed.

Aortic Aneurysm Cohort Exclusion Criteria

At the time of treatment, the patient must not have met any of the following criteria:

1. Patient required emergency surgery due to aneurysm rupture.

Dialysis Access Cohort Exclusion Criteria

At the time of treatment, the patient must not have met any of the following criteria:

1. The patient had a previous documented and unsuccessfully treated ipsilateral central venous stenosis via imaging technique.
2. The patient was taking maintenance immunosuppressant medication at the time of implant such as rapamycin, mycophenolate or mycophenolic acid, prednisone (> 10 mg), cyclosporine, tacrolimus, or cyclophosphamide.
3. The patient has had a previous instance of Heparin-Induced Thrombocytopenia type 2 (HIT-2) or has known sensitivity to heparin.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of three cohorts. Patients that have had treatment with GORE-TEX® Vascular Grafts or GORE® PROPATEN® Vascular Graft for PAD, aortic aneurysms, or dialysis access are eligible for consideration for enrollment in the registry.
  Patients will be selected from hospital database.
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- France (3):
  - Centre Hospitalier Unversitaire d'Angers, Angers
  - CHRU de Besançon, Besançon
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Italy (3):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, SOC Chirurgia Vascolare, Ancona
  - Unità di Chirurgia Vascolare Ospedale San Raffaele, Milan
  - Chirurgia Vascolare Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Spain (2):
  - Hospital del Mar, Barcelona
  - Hospital Clínico Universitario San Cecilio, Granada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PAD Cohort | AAA Cohort | Dialysis Access Cohort
Started | 145 | 65 | 146
Completed | 45 | 52 | 72
Not Completed | 100 | 13 | 74

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAD Cohort | AAA Cohort | Dialysis Access Cohort | Total
Number analyzed (Participants) | 145 | 65 | 146 | 356
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 25 | 55 | 112
  >=65 years | 113 | 40 | 91 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (10.7) | 65.9 (7.06) | 66.5 (13.1) | 68.7 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 8 | 68 | 115
  Male | 106 | 57 | 78 | 241
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 46 | 0 | 54 | 100
  France | 96 | 65 | 36 | 197
  Spain | 3 | 0 | 56 | 59

OUTCOME MEASURES:

1. Primary Outcome: PAD Cohort: Primary Safety Outcome: Device-related Seroma or Infection
Description: Clinical evidence of an infectious process in the direct vicinity of the access site or distal to the treated vascular site or seroma classified by the registry investigator as primarily related to the registry device.
Time Frame: Data were collected retrospectively from health registries, for up to 5 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 0 [0 to 0]

2. Primary Outcome: PAD Cohort: Primary Performance Outcome: Secondary Patency (Revascularization)
Description: Patency of the study graft with additional or secondary surgical or endovascular procedures to restore flow to the graft after occlusion or stenosis of the graft or its anastomoses.
  The only exceptions that do not disqualify the graft for secondary patency are procedures performed for disease beyond the graft and its two anastomoses.
Time Frame: Data were collected retrospectively from health registries, for up to 5 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 75.4 [66.3 to 82.4]

3. Primary Outcome: Aortic Aneurysm Cohort: Primary Safety Outcome: Survival Through 5 Years
Description: All Cause survival
Time Frame: Data were collected retrospectively from health registries, for up to 5 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AAA Cohort
Number analyzed (Participants) | 65
percentage of participants | 81.3 [69.4 to 88.9]

4. Primary Outcome: Aortic Aneurysm Cohort: Primary Performance Outcome: Primary Patency Through 5 Years
Description: Patency of the study graft without additional or secondary surgical or endovascular procedures to maintain or restore flow to the graft. The only exceptions that do not disqualify the graft for primary patency are procedures performed for disease beyond the graft and its two anastomoses.
Time Frame: Data were collected retrospectively from health registries, for up to 5 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AAA Cohort
Number analyzed (Participants) | 65
percentage of participants | 96.7 [87.3 to 99.2]

5. Primary Outcome: Dialysis Access Cohort: Primary Safety Outcome: Device-related Infection Through 2 Years
Description: Clinical evidence of an infectious process in the direct vicinity of the access site classified by the study investigator as primarily related to the study device.
Time Frame: Data were collected retrospectively from health registries, for up to 2 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dialysis Access Cohort
Number analyzed (Participants) | 146
percentage of participants | 0 [0 to 0]

6. Primary Outcome: Dialysis Access Cohort: Useable Access Circuit (Reported as Secondary Patency) Through 2 Years
Description: Patency of the study graft from the time of access creation or placement until access abandonment.
Time Frame: Data were collected retrospectively from health registries, for up to 2 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dialysis Access Cohort
Number analyzed (Participants) | 146
percentage of participants | 74.3 [65.7 to 81.0]

7. Secondary Outcome: Peripheral Artery Disease Cohort: Limb Salvage Through 1 Year
Description: Freedom from an amputation above the level of the ankle of the index limb
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 98.3 [93.3 to 99.6]

8. Secondary Outcome: Peripheral Artery Disease Cohort: Amputation-free Survival Through 1 Year
Description: Freedom from an amputation above the level of the ankle of the index limb or all cause death
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 81.6 [73.8 to 87.3]

9. Secondary Outcome: Peripheral Artery Disease Cohort: Device-related Adverse Events Through 1 Year
Description: Any untoward medical occurrence classified by the registry investigator as primarily related to the registry device
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 0 [0 to 0]

10. Secondary Outcome: Peripheral Artery Disease Cohort: Primary Patency Through 1 Year
Description: as for outcome 4
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 73.4 [64.9 to 80.1]

11. Secondary Outcome: Peripheral Artery Disease Cohort: Device-related Infection Requiring Reoperation Through 5 Years
Description: Clinical evidence of an infectious process in the direct vicinity of the access site or distal to the treated vascular site classified by the registry investigator as primarily related to the registry device and required surgical intervention
Time Frame: Data were collected retrospectively from health registries, for up to 5 years after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAD Cohort
Number analyzed (Participants) | 145
percentage of participants | 0 [0 to 0]

12. Secondary Outcome: Dialysis Access Cohort: Primary Patency Through 1 Year
Description: Interval following intervention until the next access thrombosis or repeated intervention.
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dialysis Access Cohort
Number analyzed (Participants) | 146
percentage of participants | 60.8 [52.0 to 68.4]

13. Secondary Outcome: Dialysis Access Cohort: Device-related Adverse Events Through 1 Year
Description: Any untoward medical occurrence classified by the registry investigator as primarily related to the registry device
Time Frame: Data were collected retrospectively from health registries, for up to 1 year after index procedure date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dialysis Access Cohort
Number analyzed (Participants) | 146
percentage of participants | 6.3 [3.2 to 12.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected retrospectively from health registries, for up to 5 years after index procedure date
Arm/Group | PAD Cohort | AAA Cohort | Dialysis Access Cohort
All-Cause Mortality (participants affected / at risk) | 54/145 | 12/65 | 27/146
Serious Adverse Events (participants affected / at risk) | 130/145 | 50/65 | 101/146
Other Adverse Events (participants affected / at risk) | 8/145 | 11/65 | 12/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAD Cohort (N=145) | AAA Cohort (N=65) | Dialysis Access Cohort (N=146)
Acute anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Acute heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block third degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Cardio-respiratory failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease progression (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decompensated heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Decompensation cardiac (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Heart attack (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 4 (5) | 0 (0) | 1 (1)
Left cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple vessel coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0)
Non ST segment elevation acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Silent myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Polycystic hepatorenal disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Multinodular goiter (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Digestion impaired (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epigastric hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage of digestive tract (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage intraabdominal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage of digestive tract (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Intestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Jejunal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mesenteric ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sessile colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Superior mesenteric artery dissection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Calf swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical condition decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Groin swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma injection site (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site hematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site seroma (General disorders) | 2 (2) | 0 (0) | 0 (0)
In-stent venous stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Multiple organ failure (General disorders) | 1 (1) | 3 (3) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Reduced general condition (General disorders) | 1 (1) | 1 (1) | 0 (0)
Stent stenosis (General disorders) | 2 (2) | 0 (0) | 3 (3)
Stent thrombosis (General disorders) | 4 (8) | 2 (3) | 12 (13)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Unknown cause of death (General disorders) | 12 (12) | 1 (1) | 3 (3)
Upper limb oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular stent-graft stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Walking difficulty (General disorders) | 0 (0) | 1 (1) | 0 (0)
Wound healing delayed (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculous cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess on buttock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Arteriovenous graft site infection (Infections and infestations) | 4 (5) | 0 (0) | 3 (3)
Aspiration pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Epididymo-orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epiduritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Foot abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene toe (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Inguinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis of the foot (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pilonidal sinus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Pseudoaneurysm infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Purulent discharge (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Renal cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Schistosomiasis bladder (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (6) | 0 (0) | 2 (2)
Septic arthritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Septicemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Surgical site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Surgical wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular graft infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Vascular stent infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Achilles tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acute subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Arteriovenous fistula site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Arteriovenous fistula site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula site stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 13 (20)
Arteriovenous graft site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion of knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
False aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture vertebral (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fractured thumb (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Incision site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Incision site hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration of face (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar spine compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural bleeding (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound necrosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Surgical wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Trochanteric femoral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site bleeding (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular access site necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 25 (36)
Vascular access steal syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 6 (7) | 2 (2) | 5 (6)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pedal pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperosmolar hyperglycaemic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Water retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hips osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in toe (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Antral carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bone metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon adenomatous polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colonic tubular adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Esophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Kidney tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumor compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Amputation stump pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cognitive impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cruralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Internal carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Syncopal attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Unilateral carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 12 (15) | 0 (0) | 9 (15)
Stent occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 22 (33) | 0 (0) | 3 (3)
Anxiety depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 3 (3) | 2 (2) | 3 (3)
Acute renal insufficiency (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Chronic renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure aggravated (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal insufficiency aggravated (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory decompensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Basilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Blistering (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bullous pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Below knee amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Transmetatarsal amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Abdominal aortic aneurysm hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute limb ischaemia (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Acute limb ischemia (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Aneurysm thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 2 (4) | 0 (0) | 0 (0)
Chronic limb ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic limb-threatening ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Critical limb ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Critical limb ischemia (Vascular disorders) | 10 (14) | 1 (1) | 0 (0)
Cyanosis peripheral (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Digital necrosis (Vascular disorders) | 4 (4) | 0 (0) | 1 (1)
External iliac artery stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral artery stenosis (Vascular disorders) | 5 (7) | 0 (0) | 0 (0)
Groin hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Hemorrhagic shock (Vascular disorders) | 1 (1) | 4 (4) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Ischemic limb pain (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Leg ischemia (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lower limb ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lower limb ischemia (Vascular disorders) | 4 (6) | 3 (4) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vein stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Popliteal artery aneurysm (Vascular disorders) | 2 (2) | 1 (2) | 0 (0)
Popliteal artery aneurysm enlargement (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 0 (0) | 5 (5)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial femoral artery occlusion (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Type A aortic dissection (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Type B aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Uncontrolled hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous bleeding (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAD Cohort (N=145) | AAA Cohort (N=65) | Dialysis Access Cohort (N=146)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 12 (15)
Anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT05124184/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05124184/SAP_001.pdf